CLINICAL TRIAL: NCT05115812
Title: Renal Autotransplantation; Case Series
Status: Enrolling by invitation | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 025.HPB.2021.D
Record Dates: First submitted 2021-10-08; First posted 2021-11-10 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Renal Vascular Disease; Nutcracker Syndrome, Renal; Pelvic Trauma; Loin Pain-Hematuria Syndrome; Renal Tumor; Congestion, Venous
MeSH Terms: conditions — Renal Nutcracker Syndrome; Carcinoma, Renal Cell; Hyperemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RAT: patients having undergone robotic-assisted RAT procedure
  Interventions: Procedure: Pre-Operative Information; Procedure: Intra-Operative Data; Other: Post-Operative Data (up to discharge); Other: Short-Term Follow-Up Data

INTERVENTIONS:
Procedure: Pre-Operative Information — Demographics (e.g., age, gender), patient characteristics (e.g., BMI, American Society of Anesthesiologists class), and pre-operative medical history (e.g., tobacco use; comorbidities: hypertension, cardiopulmonary disease, diabetes; indication for RAT; lesions; previous renal revascularization; serum creatinine level).
Procedure: Intra-Operative Data — Operative time, total OR time, concomitant procedures, transfusions, conversions, intraoperative adverse events, autotransplantation technique
Other: Post-Operative Data (up to discharge) — Postoperative adverse events, discharge status, hospital length of stay, information on enhanced recovery program
Other: Short-Term Follow-Up Data — Adverse events, re- admissions, re-operations related to the index procedure

SUMMARY:
Renal autotransplantation (RAT) is a method of removing a kidney from its place of origin in a patient, repairing it, and transplanting it in another location of the body, generally the iliac fossa of the same patient.RAT is a relatively new technique; the first ever RAT procedure in the US was performed in 1963. Advances in preservation and transplantation techniques have made RAT a modality that can be utilized in complex renal diseases. RAT is indicated for conditions such as renal vascular disease, nutcracker syndrome, pelvic venous congestion, pelvic trauma, refractory stone disease and, in some cases, loin pain hematuria syndrome and conventionally unresectable renal tumors.

Irrespective of the excellent outcomes shown by RAT, the conventional open approach requires a large midline xiphoid-to-pubis or flank incision for donor nephrectomy with a second pelvic incision for renal transplantation into the iliac fossa.The current gold standard approach to RAT is a laparoscopic nephrectomy followed by open auto-transplantation. However, this approach still requires a large pelvic incision. Robotic technology enables us to perform more complex minimally invasive surgery. Gordon et al. performed and reported the first completely intracorporeal robotic RAT to repair a ureteral injury in 2014.

DETAILED DESCRIPTION:
This is a retrospective chart review case series study of all consecutive cases in which robotic RAT was performed that meet the study inclusion and exclusion criteria. The case series will be performed starting from January 2018 until June 2021 to include all cases of robotic RAT procedures.

Perioperative and short-term clinical data will be obtained from the EMR. All the data variables will be documented in the case report forms.

Because the data will have been de-identified and is archival in nature, there will be no active subject recruitment and no patient consenting is required.

ELIGIBILITY:
Inclusion Criteria:

* Subject was 18 years or older at the time of the procedure
* Subject who has undergone robotic RAT irrespective of the underlying etiology.

Exclusion Criteria:

* Subjects who do not meet the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective chart review case series study of all consecutive cases in which robotic RAT was performed that meet the study inclusion and exclusion criteria. The case series will be performed starting from January 2018 until June 2021 to include all cases of robotic RAT procedures.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Baseline patient characteristics | January 2018 until June 2021
  Demographics-age
Baseline patient characteristics- BMI | January 2018 until June 2021
  BMI, based on the American Society of Anesthesiologists status classification
Baseline patient characteristics- Tobacco use | January 2018 until June 2021
  Medical History: tobacco use
Baseline patient characteristics- Gender | January 2018 until June 2021
  Demographics: gender
Baseline patient characteristics- Hypertension | January 2018 until June 2021
  Medical History: hypertension
Baseline patient characteristics- Diabetes | January 2018 until June 2021
  Medical History: diabetes
Baseline patient characteristics-cardiopulmonary disease | January 2018 until June 2021
  Medical History: cardiopulmonary disease
Baseline patient characteristics-indication for RAT (Renal Autotransplantation | January 2018 until June 2021
  Medical History: indication for RAT (Renal Autotransplantation)
Baseline patient characteristics-lesions | January 2018 until June 2021
  Medical History: lesions
Baseline patient characteristics-previous renal revascularization | January 2018 until June 2021
  Medical History: previous renal revascularization
Baseline patient characteristics-serum creatinine level | January 2018 until June 2021
  Medical History: serum creatinine level
short-term clinical data-Adverse events, | up to 30 days post discharge
  Adverse events, re- admissions, re-operations related to the index procedure
intraoperative characteristics-Operative time | January 2018 until June 2021
  Operative time
intraoperative characteristics-total OR time | January 2018 until June 2021
  total OR time
intraoperative characteristics-concomitant procedures | January 2018 until June 2021
  concomitant procedures
intraoperative characteristics-transfusions | January 2018 until June 2021
  transfusions
intraoperative characteristics-conversions | January 2018 until June 2021
  conversions
intraoperative characteristics-intraoperative adverse events | January 2018 until June 2021
  intraoperative adverse events
intraoperative characteristics-autotransplantation technique | January 2018 until June 2021
  autotransplantation technique
post-operative characteristics-Post-operative adverse events | January 2018 until June 2021
  Post-operative adverse events
post-operative characteristics-discharge status | January 2018 until June 2021
  discharge status
post-operative characteristics-hospital length of stay | January 2018 until June 2021
  hospital length of stay
post-operative characteristics-information on enhanced recovery program | January 2018 until June 2021
  information on enhanced recovery program

CONTACTS AND LOCATIONS:
Locations (1):
- Liver Institute of Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No